CLINICAL TRIAL: NCT00757224
Title: Parental Education on Passive Smoke Exposure and Respiratory Diseases in Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Arnon Elizur, MD, The institute of allergy and pulmonary medicine, Asaf Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 147/08
Record Dates: First submitted 2008-09-21; First posted 2008-09-23 (Estimated); Last update posted 2008-09-23 (Estimated); Status verified 2008-09

CONDITIONS: Tobacco Smoke Pollution
MeSH Terms: interventions — Counseling

ARMS (3):
- non-smoking (No Intervention)
- smoking parents A (No Intervention)
- smoking parents B (Experimental): Parents will be educated on the hazards of passive smoke exposure and ways to reduce it
  Interventions: Behavioral: Guidance

INTERVENTIONS:
Behavioral: Guidance — Smoking parents will receive education on the association between parental smoking and respiratory morbidity in the infant. They will also be offered ways to reduce smoke exposure of their infants.
  Arms: smoking parents B

SUMMARY:
Parental smoking is associated with increased frequency of respiratory diseases including hospitalizations in infants.

Study hypothesis: Parental education regarding the association between parental smoking and respiratory diseases in the infant, and guidance on ways to decrease smoke exposure by the infant, provided shortly after the infant is born, will decrease infants' morbidity.

DETAILED DESCRIPTION:
Mothers who are in Maternity ward following birth will fill a questionnaire regarding smoking habits. Parents will be divided into non-smokers and smokers. Half of the smoking mothers will receive guidance regarding the association between parents smoking and respiratory diseases in the infant. They will also get ideas on how to reduce smoke exposure by their infant. 3 months and 1 year later all parents will be contacted by phone and asked about their children's health.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at Asaf Harofeh Medical Center
* Infants born at >35W gestational age

Exclusion Criteria:

* Infants requiring any supportive treatment (supplemental O2, fluids, glucose, antibiotics)

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2008-10; Primary Completion 2008-11 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
The number of episodes of cough/wheeze/asthma/bronchitis during the first 3 months and 1 year. | 3 months and 1 year

SECONDARY OUTCOMES:
The number of ED visits and hospitalizations for respiratory diseases in the first 3 months and 1 year | 3 months and 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Asaf Harofeh Medical Center, Ẕerifin, Israel